CLINICAL TRIAL: NCT03941236
Title: An Extension Trial Evaluating the Long-term Safety and Efficacy of Dasiglucagon for the Treatment of Children With Congenital Hyperinsulinism
Brief Title: Extension Trial Evaluating the Long-term Safety and Efficacy of Dasiglucagon in Children With Congenital Hyperinsulinism
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZP4207-17106
Record Dates: First submitted 2019-05-02; First posted 2019-05-07 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Congenital Hyperinsulinism
MeSH Terms: conditions — Congenital Hyperinsulinism | interventions — dasiglucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dasiglucagon open-label (Experimental): Dasiglucagon treatment as an SC infusion in the dose range 10-70 μg/h titrated individually +/- standard of care
  Interventions: Drug: dasiglucagon

INTERVENTIONS:
Drug: dasiglucagon — Glucagon analog
  Other Names: ZP4207

SUMMARY:
This is an open-label, multinational, multicenter, long-term safety and efficacy extension trial in patients with Congenital Hyperinsulinism (CHI) who completed either ZP4207-17103 or ZP4207-17109 (defined as lead-in trials).

The primary objective is to evaluate the long-term safety of dasiglucagon administered as a subcutaneous (SC) infusion in children with CHI.

ELIGIBILITY:
Inclusion Criteria:

* Completed treatment in either Trial ZP4207-17103 or ZP4207-17109
* Expected to continue to have a positive benefit-risk assessment for treatment with dasiglucagon (based on considerations of glycemic effect, tolerability, and nature and frequency of adverse events experienced in the lead-in trial)

Exclusion Criteria:

* The patient developed any conditions prohibited by the lead-in trial, requires medication prohibited by the lead-in trial, or has other new complications that preclude participation in the investigator's opinion.

Ages: 5 Weeks to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Baseline through treatment completion, up to 3 years
  Number of adverse events occurring up to Month 1, Month 1 to Month 3 and in each 3-month period for the first year; subsequent years will have longer periods assigned for analysis

SECONDARY OUTCOMES:
Amount of gastric carbohydrates administered to treat hypoglycemia | Baseline through treatment completion, up to 3 years
  Total amount of gastric carbohydrates administered via nasogastric tube or gastrostomy per week to treat hypoglycemia
Nasogastric (NG) tube or gastrostomy removal | Baseline through treatment completion, up to 3 years
  Time to removal of NG tube or gastrostomy
Pancreatic surgery | Baseline through treatment completion, up to 3 years
  Time to pancreatic surgery (sub-total or total pancreatectomy)
Time in hypoglycemia | Baseline through treatment completion, up to 3 years
  Continuous glucose monitoring (CGM) percent time <70 mg/dL (3.9 mmol/L)
Hypoglycemia episodes | Baseline through treatment completion, up to 3 years
  Rate of CGM-detected hypoglycemia episodes <70 mg/dL (3.9 mmol/L) for 15 minutes or more
Clinically significant episodes of hypoglycemia | Baseline through treatment completion, up to 3 years
  Rate of clinically significant CGM-detected hypoglycemia episodes <54 mg/dL (3.0 mmol/L) for 15 minutes or more
Gastric carbohydrate administrations | Baseline through treatment completion, up to 3 years
  Number of gastric carbohydrate administrations (nasogastric tube or gastrostomy) to treat hypoglycemia
Nightly gastric carbohydrate administrations | Baseline through treatment completion, up to 3 years
  Number of nightly (midnight to 6 am) gastric carbohydrate administrations (nasogastric tube or gastrostomy) to treat hypoglycemia
Extent of hypoglycemia | Baseline through treatment completion, up to 3 years
  Extent of hypoglycemia (area over the glucose curve [AOCglucose] below 70 mg/dL [3.9 mmol/L]) as measured by continous glucose monitoring (CGM)
Extent of clinically significant hypoglycemia | Baseline through treatment completion, up to 3 years
  Extent of hypoglycemia (area over the glucose curve [AOCglucose] below 54 mg/dL [3.0 mmol/L]) as measured by continous glucose monitoring (CGM)
Diazoxide dose | Baseline through treatment completion, up to 3 years
  Reduction in diazoxide dose in mg/kg body weight/day from start of lead-in trial
Somatostatin analog dose | Baseline through treatment completion, up to 3 years
  Reduction in somatostatin analog dose from start of lead-in trial
Prescribed amount of continuous gastric carbohydrate administration | Baseline through treatment completion, up to 3 years
  Change in total amount of prescribed continuous gastric carbohydrate administration from start of lead-in trial (g/day)
Prescribed duration of continuous gastric carbohydrate administration | Baseline through treatment completion, up to 3 years
  Change in prescribed duration of infusion of continuous gastric carbohydrate administration from start of lead-in trial (h/day)
Prescribed duration of nightly continuous gastric carbohydrate administration | Baseline through treatment completion, up to 3 years
  Change in prescribed duration of infusion of nightly (8 pm - 8 am) continuous gastric carbohydrate administration from start of lead-in trial (h/day)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Information Desk, Study Director — Zealand Pharma
Locations (10):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Endocrinology and Diabetes Clinic, Fort Worth, Texas
- Germany (2):
  - University Hospital Düsseldorf, Department of Pediatrics, Düsseldorf
  - Otto von Guericke University Magdeburg, Department of Pediatrics, Magdeburg
- Hadassah Medical Center, Jerusalem, Israel
- United Kingdom (4):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Alder Hey Children's Hospital NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03941236/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT03941236/SAP_001.pdf